CLINICAL TRIAL: NCT02012244
Title: Effects of Postoperative Pain Management on Immune Function After Laparoscopic Resection of Colorectal Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Severance Hospital (Other)
Responsible Party: Principal Investigator, So Yeon Kim, Assistant professor, Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 4-2013-0044
Record Dates: First submitted 2013-12-07; First posted 2013-12-16 (Estimated); Last update posted 2016-01-12 (Estimated); Status verified 2016-01

CONDITIONS: Colorectal Surgery
Keywords: analgesia; colorectal surgery; immunity; local anesthetics; opioids
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- fentanyl-based analgesia (Experimental): fentanyl intravenous patient-controlled analgesia + additional pethidine
  Interventions: Drug: fentanyl-based analgesia
- local anesthetic wound infiltration-based anlagesia (Experimental): continuous wound inflitration with ropivacaine + tramadol intravenous patient-controlled analgesia + additional ketorolac or propacetamol
  Interventions: Drug: local anesthetic wound infiltration-based anlagesia

INTERVENTIONS:
Drug: fentanyl-based analgesia — fentanyl based patient-controlled analgesia + additional pethidine for postoperative 48 hour
  Arms: fentanyl-based analgesia
Drug: local anesthetic wound infiltration-based anlagesia — continuous wound inflitration with ropivacaine + tramadol patient-controlled analgesia + additional ketorolac or propacetamol for postoperative 48 hour
  Arms: local anesthetic wound infiltration-based anlagesia

SUMMARY:
The purpose of this study is to compare postoperative immune function (e.g. NK cell activity) of fentanyl-based analgesic regimen versus local anesthetic wound infiltration-based anlagesic regimen after laparoscopic colorectal surgery

ELIGIBILITY:
Inclusion Criteria:

* ASA class I-III
* 20-80 years old
* elective laparoscopic colorectal surgery for cancer

Exclusion Criteria:

* drug allergy
* significant renal or hepatic impairment
* sign of infection

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
NK cell activity | 48 hours
  NK cell activity : preoperation, POD 1, POD 2
IL-2 | 48 hours
  IL-2 level : preoperation, POD 1, POD 2

SECONDARY OUTCOMES:
Complication and recurrence | 1 year
  Postoperative complication, recurrence

OTHER OUTCOMES:
Inflammatory responses | 48 hours
  White blood cell, neutrophil, C-reactive protein (CRP) : preoperation, POD 1, POD 2

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine and Anesthesia and Pain Research Institute, Yonsei University College of Medicine, Sedoul, South Korea